CLINICAL TRIAL: NCT02293187
Title: The Impact of Supplemental Vitamin D on Serum 25-hydroxyvitamin D Levels and Short Term Indicators of Physical Function
Brief Title: Impact of Vitamin D on 25-hydroxyvitamin D Levels and Physical Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Bess Dawson-Hughes, Director, Bone Metabolism Laboratory, HNRCA, Tufts University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: 2710
Record Dates: First submitted 2014-07-23; First posted 2014-11-18 (Estimated); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Vitamin D Deficiency; Sarcopenia
Keywords: vitamin D; muscle performance; falls
MeSH Terms: conditions — Vitamin D Deficiency; Sarcopenia | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- vitamin D3 (Active Comparator): Vitamin D3, 800 IU will be given initially; after 4 months if D level < 70 nmol/L, increase dose to 1600 IU for remainder of study.
  Interventions: Dietary Supplement: vitamin D3
- Placebo (Placebo Comparator): Placebo, microcrystalline cellulose
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: vitamin D3 — Dose for intervention arm is 800 IU/day for first 4 months. At 4 months, if vitamin D level <70 nmol/L, a second 800 IU capsule will be added to regimen (total of 1600 IU/d) for remainder of study.
  Other Names: cholecalciferol
  Arms: vitamin D3
Other: Placebo — Those in the placebo group will receive 1 capsule for first 4 months. At 4 month visit, one capsule will be added to regimen to be taken throughout the remainder of the study.
  Other Names: microcystalline cellulose
  Arms: Placebo

SUMMARY:
This one-year study will test the hypothesis that supplementation with vitamin D will improve lower extremity muscle performance in older men and women with vitamin D insufficiency.

DETAILED DESCRIPTION:
Vitamin D may have favorable effects on muscle but evidence is mixed. It appears that subjects with low starting levels of 25-hydroxyvitamin D (25OHD) who receive adequate doses of vitamin D are the most likely to benefit. Vitamin D supplements are being widely recommended, however the amount of vitamin D needed to achieve the desired level of 25-hydroxyvitamin D in the circulation varies widely among individuals. In this randomized, placebo-controlled trial, we will determine whether treating older adults with low starting 25OHD levels for one year with up to 1600 IU per day of vitamin D3 will improve muscle performance (e.g., lower extremity muscle power) and reduce muscle wasting (defined as reducing nitrogen excretion). Subjects in the vitamin D group will initially take 800 IU of vitamin D3 daily. If they have not achieved the desired level of 70 nmol/L after 4 mo, their dose will be doubled to 1600 IU per day for the remainder of the one-year study. The maximal dose of vitamin D3 to be taken in this study,1600 IU per day, is lower than the current safe upper limit of 4,000 IU per day set by the Institute of Medicine. Up to 100 healthy men and women, age 60 years and older will participate in this study. This investigation should increase our understanding of the impact of supplemental vitamin D on muscle performance.

ELIGIBILITY:
Inclusion Criteria:

* Men and postmenopausal women age 60 years and older
* Women must be at least 1 year since last menses.
* Subjects must agree not to take their own vitamin D in amounts >600 IU/day (for ages 51-70 years) or >800 IU/day (for ages 71 - 80 years) or more than 600 mg/day of supplemental calcium.
* Subjects must agree not to have had more than 30 minutes/day of sun exposure at a southern latitude (< 34 degrees N) in the 2-month period prior to screening and not to travel south and be exposed to sunshine in the 3-month period prior to their final visit.
* They will agree not to use tanning salons during the study.
* Screening serum 25OHD of 20 to 50 nmol/L (8.0 to 20 ng/ml).

Exclusion Criteria:

* Kidney stones - in the last 3 years
* Calculated glomerular filtration rate < 30 ml/min
* Screening fasting spot urinary calcium:creatinine ratio (Ca:Cr) > 0.325 (corresponding to a 24-hr urine calcium of 350 mg)
* Serum calcium exceeding upper normal limit (reference range 8.3 -10.2 mg/dl)
* Other abnormalities in screening labs, at the discretion of the study physician (PI)
* Sarcoidosis
* Evidence of chronic liver disease, including alcoholism
* Cancer treatment in the last year (except basal cell carcinoma) or terminal illness
* Treatment in the last 6 months with estrogen, raloxifene, calcitonin, or testosterone (vaginal estrogen use okay)
* High dose thiazide therapy (>37.5 mg).
* Treatment in the last year with teriparatide or denosumab
* Treatment in the lsat 2 years with bisphosphonates
* Oral corticosteroid therapy for over 3 weeks within the last 6 months
* Anticonvulsant therapy
* Physical conditions such as osteoarthritis, rheumatoid arthritis, heart failure or hemiplegia severe enough to prevent reasonable physical activity.
* Non-English speaking subjects (We can't be confident that non-English speaking subjects could accurately identify intakes of calcium and vitamin D from non-study sources and this could increase their risk of toxicity from study drug.
* Other abnormalities in screening labs, at the discretion of the study physician (the PI)

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-03-23 (Actual); Primary Completion 2017-09-13 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
The effect of supplemental vitamin D3 vs placebo on leg power and nitrogen excretion. | 12 months
  Aim of the study is to look at the effect of supplemental vitamin D3 vs placebo on leg power and nitrogen excretion.To determine Vitamin D will improve leg power and reduce muscle wasting, as measured by 24-hr nitrogen excretion.

SECONDARY OUTCOMES:
To describe the safety (assessed by serum calcium) of the administered doses of vitamin D3. | 12 months
  To describe the safety (assessed by serum calcium) of the administered doses of vitamin D3.

OTHER OUTCOMES:
To determine the effect of supplemental vitamin D3 vs placebo on SPPB. | 12 months
  To determine the effect of supplemental vitamin D3 vs placebo on SPPB.
To determine the effect of supplemental vitamin D3 vs placebo on handgrip. | 12 months
  To determine the effect of supplemental vitamin D3 vs placebo on handgrip.
To determine the effect of supplemental vitamin D3 vs placebo on stair climb. | 12 months
  To determine the effect of supplemental vitamin D3 vs placebo on stair climb.
To determine the effect of supplemental vitamin D3 vs placebo on backward walking. | 12 months
  To determine the effect of supplemental vitamin D3 vs placebo on backward walking.

CONTACTS AND LOCATIONS:
Overall Officials: Bess Dawson-Hughes, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Jean Mayer USDA Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shea MK, Fielding RA, Dawson-Hughes B. The effect of vitamin D supplementation on lower-extremity power and function in older adults: a randomized controlled trial. Am J Clin Nutr. 2019 Feb 1;109(2):369-379. doi: 10.1093/ajcn/nqy290. PMID 30715090